CLINICAL TRIAL: NCT02346292
Title: Observational Multicenter Non-interventional Study on COPD Patients Treatment Strategies at the Time of Hospital Discharge and Within 12 Months of Follow-up on an Outpatient Primary Care Basement
Acronym: CLOUD
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RRU-XXX-2014/1
Record Dates: First submitted 2015-01-14; First posted 2015-01-27 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: COPD
Keywords: COPD; Spirometry; severe and very severe COPD; COPD exacerbations; therapy schemes; therapy changes
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients of both genders aged 40 years and older, smokers, with smoking history more than 10 pack-years, with severe and very severe COPD who were hospitalized with COPD exacerbation

SUMMARY:
The study is an observational multicenter descriptive study. It is planned to enroll approximately 1250 subjects with severe and very severe COPD hospitalized for the reason of COPD exacerbation into departments of pulmonology or therapy. The study will be conducted in approximately 20-25 institutions of treatment and prevention in Russian Federation and will include about 50 to 60 subject at each clinical site.

DETAILED DESCRIPTION:
The study is an observational multicenter descriptive study. It is planned to enroll approximately 1000 subjects with severe and very severe COPD hospitalized for the reason of COPD exacerbation into departments of pulmonology or therapy. The study will be conducted in approximately 20-25 institutions of treatment and prevention in Russian Federation and will include about 50 to 60 subject at each clinical site.

This is an observational study, so there is no treatment protocol or subjects' management recommendations required. The study subjects receive medical treatment according to the routine practice for their disease in Russian Federation. A subject's participation in this clinical study should not affect character and amount of care provided according to the routine clinical practice.

The study includes 5 clinical visits: Study Enrolment Visit, Month 3 Visit, Month 6 visit, Month 9 Visit, Month 12 visit / End of Study Visit.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent . Men and women at least 40 years old, with smoking history more than 10 pack-years.
* Hospitalization for the reason of COPD exacerbation (exacerbation defined as acute condition, different from typical fluctuations of general condition and requiring change of therapy).
* Diagnosis of severe or very severe COPD based on final spirometry (performed in a standardized manner using salbutamol 400 mg), or history of diagnosis of severe or very severe COPD based on spirometry performed during 6 months before the hospitalization.

Exclusion Criteria:

* Participation in any interventional study.
* Concomitant respiratory diseases, i.e. confirmed or suspected malignancy or any other serious condition, including lung tumor, lung fibrosis, interstitial lung disease, tuberculosis, sarcoidosis.
* Patient is unable or unwilling to complete questionnaires, unable to understand study procedures, or other reasons which, in the investigator's opinion, could affect study procedures performance.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both genders aged 40 years and older, smokers, with smoking history more than 10 pack-years, with severe and very severe COPD who were hospitalized with COPD exacerbation
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2015-03-31 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with severe and very severe COPD who received prescription of therapy, including different schemes of inhaled glucocorticoids use, according to main principles of COPD therapy (GOLD 2014 recommendations) | up to 12 months

SECONDARY OUTCOMES:
Description of social characteristics (days of disability, etc.), economical status of subjects if applicable (if patient agreed) (average monthly income) with severe and very severe COPD hospitalized for the reason of COPD exacerbation | at the time of 1st visit
% of subjects with severe and very severe COPD for whom scheme of inhaled glucocorticoids use was changed after 3, 6, 9, and 12 months of follow-up (outpatient conditions after discharge from the hospital) | at the moment of discharge and after 3, 6, 9, and 12 months of follow-up
Frequency and reasons of treatment scheme correction during follow-up after its prescription at the moment of discharge from the hospital | at the moment of discharge and after 3, 6, 9, and 12 months of follow-up
  As reasons of treatment changes and/or its correction it will be measured with:
  1. Number of hospitalizations in the previous 3 months before enrollment and in 3, 6, 9, 12 months;
  2. Number or emergency calls, outpatient care settings visits in the previous 3 months before enrollment and in 3, 6, 9, 12 months;
  3. Number of exacerbations and number of related hospitalizations in the previous 3 months before enrollment and in 3, 6, 9, 12 months.
  4. Number of pneumonia cases in the previous 3 months before enrollment and in 3, 6, 9, 12 months.
% of subjects with severe and very severe COPD who during the follow-up period attended medical institution for the correction of treatment scheme prescribed at the moment of discharge from the hospital | at the moment of discharge and after 3, 6, 9, and 12 months of follow-up
% of subjects with severe and very severe COPD, received treatment with short acting anticholinergic drugs, SABA, LABA, LAMA, oral CS, FDC, phosphodiesterase type 4 inhibitors, theophylline | at the moment of discharge and after 3, 6, 9, and 12 months of follow-up
% of patients with asthma-COPD overlap syndrome among all subjects with severe and very severe COPD hospitalized for the reason of COPD exacerbation | at the time of 1st visit and 12 months of follow-up
% of subjects with asthma-COPD overlap syndrome who received treatment with inhaled glucocorticoids both | at the moment of discharge and after 3, 6, 9, and 12 months of follow-up
% of patients with severe and very severe COPD, who received treatment with short acting anticholinergic drugs, SABA, LABA, LAMA, oral CS, FDC, phosphodiesterase type 4 inhibitors, theophylline, among all subjects with ACOS | at the moment of discharge and after 3, 6, 9, and 12 months of follow-up
EQ-5D results | at the moment of discharge and after 3, 6, 9, and 12 months of follow-up
CAT results | at the moment of discharge and after 3, 6, 9, and 12 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Bedenkov, Medical Director, Study Director — AstraZeneca; Sergey Avdeev, MD, PHD, Principal Investigator — Federal State Institution "Scientific Research Institute of Pulmonology" FMBA of Russia; Andrey Belevsky, PHD, Principal Investigator — Federal State Institution "Scientific Research Institute of Pulmonology" FMBA of Russia
Locations (30):
- Russia (30):
  - Research Site, Barnaul
  - Research Site, Blagoveshchensk
  - Research Site, Chelyabinsk
  - Research Site, Cherepovets
  - Research Site, Chita
  - Research Site, Gatchina
  - Research Site, Izhevsk
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Kirov
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Kursk
  - Research Site, Moscow
  - Research Site, Naberezhnye Chelny
  - Research Site, Novokuznetsk
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Oryol
  - Research Site, Petrozavodsk
  - Research Site, Rostov-on-Don
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Seversk
  - Research Site, Smolensk
  - Research Site, Ufa
  - Research Site, Voronezh
  - Research Site, Yakutsk
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3274&filename=CLOUD_Study%20Report%20Summary_Redacted.pdf